CLINICAL TRIAL: NCT04038164
Title: Dog-Assisted Therapy for Children and Adolescents With FASD: a Randomized Controlled Pilot Study
Brief Title: Dog-Assisted Therapy for Children and Adolescents With FASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)94/2018
Record Dates: First submitted 2019-06-28; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: FASD
Keywords: FASD; animal-assisted therapy; dog-assisted therapy
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: The design was a randomized, rater-blinded, controlled pilot trial. Participants were randomly assigned either to DAT group (n=17) or Treatment as Usual (TAU control group) (n=16).
Who Masked: Outcomes Assessor
Masking Description: Rater-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dog-Assisted Therapy (DAT) and pharmacological treatment (Experimental): The DAT program comprised 12 manualized sessions and included two phases: 1) individual intervention (6 sessions) and 2) group activity (6 sessions). Patients participated in weekly sessions for about 3 months. Each session lasted 45 minutes. The groups were formed by 3-4 patients. Sessions included the participation of two certified therapy dogs, two technicians specialized in DAT and a psychologist. Participants in this group were visited by their psychiatrist in order to monitor their adherence to medications.
  Interventions: Behavioral: Dog-Assisted Therapy and pharmacological treatment
- Treatment as usual (TAU, pharmacological treatment) (Active Comparator): Participants received their usual treatment. They were visited by their psychiatrist in order to monitor their adherence and continuation on medications as prescribed. Inclusion and exclusion criteria were the same as for the experimental group. Participants in the TAU group did not receive DAT sessions.
  Interventions: Behavioral: Dog-Assisted Therapy and pharmacological treatment

INTERVENTIONS:
Behavioral: Dog-Assisted Therapy and pharmacological treatment — The investigators used the CTAC Method (Center of Dog Assisted Therapy) (E Domènec 2012).

SUMMARY:
The rationale of the present study was to evaluate the efficacy of DAT in children and adolescents with FASD in relation to its effects on social skills, internalized and externalized symptomatology and on severity of FASD symptoms. This objective was accomplished through a randomized controlled pilot study of DAT for children and adolescents with FASD.

DETAILED DESCRIPTION:
The rationale of this study was to evaluate the efficacy of Dog Assisted Therapy in children and adolescents with FASD. The investigators conducted a randomized, rater-blinded, controlled pilot trial in a cohort of 33 children and adolescents with FASD. Participants were randomly assigned either to DAT group (n=17) or Treatment as Usual (TAU control group) (n=16). The investigators evaluated changes on social skills, internalized and externalized symptomatology and on severity of FASD symptoms at pre-treatment and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with FASD between 6 and 18 years (FAS, pFAS or ARND)
* With or without comorbidities
* Stabilized doses of medication for at least 2 months before the study
* Patients with borderline IQ or mental retardation.

Exclusion Criteria:

* Patients who were not behaviorally stable
* Patients that required hospitalization, day hospital or more intensive treatments.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Social skills at 3 months | Pre-treatment (baseline) and post-treatment assessment (through study completion, at 3 months)
  Social Skills Improvement System-Parent Form (SSIS-P). is a 79 items scale (Likert scale 0 to 4) measuring social skills and problem behaviors in children and adolescents as reported by their parents. In the Social Skills domain, the subscales are communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. The Problem Behaviors domain includes internalizing and externalizing problems, bullying, hyperactivity/inattention and autism spectrum.
Change from baseline on Externalizing symptoms at 3 months | Pre-treatment (baseline) and post-treatment assessment (through study completion, at 3 months)
  Child Behavior Checklist (CBCL of Achenbach) parent version. to assess Internalizing and Externalizing Symptoms in patients between 4 and 18 years. The CBCL is a 113 item scale (Likert scale: 0-2) which assesses withdrawn symptoms, somatic complains, anxiety/depressive symptoms, thought problems, ADHD features, oppositional behavior and behavioral problems. Higher scores indicate more conduct problems.
Change from baseline FASD severity at 3 months | Pre-treatment (baseline) and post-treatment assessment (through study completion, at 3 months)
  Clinical Global Impression Scale for Severity(CGI-S Clinician). The Clinical Global Impression Scale for Severity (CGI-S): is a 7-point scale (1 = normal or not ill, and 7 = extremely ill) .

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vidal, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Vall d'Hebron Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vidal R, Vidal L, Lugo J, Ristol F, Domenec E, Casas T, Veiga A, Vico C, Ramos-Quiroga JA, Gomez-Barros N. Dog-Assisted Therapy vs Relaxation for Children and Adolescents with Fetal Alcohol Spectrum Disorder: A Randomized Controlled Study. J Autism Dev Disord. 2024 Aug;54(8):3133-3141. doi: 10.1007/s10803-023-06023-5. Epub 2023 Jun 20. PMID 37340213
- [Derived] Vidal R, Vidal L, Ristol F, Domenec E, Segu M, Vico C, Gomez-Barros N, Ramos-Quiroga JA. Dog-Assisted Therapy for Children and Adolescents With Fetal Alcohol Spectrum Disorders a Randomized Controlled Pilot Study. Front Psychol. 2020 May 26;11:1080. doi: 10.3389/fpsyg.2020.01080. eCollection 2020. PMID 32528389